CLINICAL TRIAL: NCT01955811
Title: Bicentric Clinical Trial With in Vitro Experiments to Assess the Effect of Fibrinogen (FGTW) on Coagulation in Thrombocytopenia
Brief Title: Study to Reveal if Fibrinogen Treatment Effects Blood Clotting Better Than a Platelet Transfusion
Acronym: FiT2012
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Dietmar Fries, M.D., Ao. Univ.-Prof. Dr., Medical University Innsbruck
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: FiT2012
Record Dates: First submitted 2013-09-02; First posted 2013-10-08 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Blood Platelet Transfusion; Blood Clotting
Keywords: platelet transfusion; Fibrinogen; blood coagulation; Thrombocytopenia; in-vitro experiments; FGTW; Fit2012; factor I; Fibrin
MeSH Terms: conditions — Thrombosis; Thrombocytopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Platelet concentrate transfusion and Human Fibrinogen (Other): Blood samples will be collected directly before the start of transfusion and 1 hour after the end of transfusion. These samples will be spiked with Human Fibrinogen and clotting tests will be performed. After 24 h after end of transfusion a clotting test will be performed again.
  Interventions: Drug: Administration of platelet concentrate and taking blood samples

INTERVENTIONS:
Drug: Administration of platelet concentrate and taking blood samples — Patient with the need of a platelet transfusion, will have 4 intervention points. 1. directly before the start of the transfusion a blood sample will be drawn. 2. Patient receives the platelet transfusion. 3. One hour after the end of transfusion a second blood sample will be drawn. 4. 24 h after the end of the platelet transfusion a further bloos sample will be collected. The first two samples will be (beside blood cell counts) spiked in-vitro with different amounts of Human fibrinogen and blood clotting tests will be performed. The same with the 3. blood sample, but without spiking steps.

SUMMARY:
Patients with need of platelet transfusion for any reason will participate in this study. Directly before the start of infusion and one hour after the end of platelet transfusion blood samples will be drawn and treated with different concentrations of Fibrinogen (a blood clotting factor) in-vitro. Blood samples with and without Fibrinogen/platelet transfusion will be compared. The study hypothesis is that treatment with Fibrinogen results in a better stabilisation of blood coagulation.

DETAILED DESCRIPTION:
In total 300 patients with the need of platelet transfusion for whatever reason will be included when meeting the inclusion- and exclusion criteria.

For all patients three visits are planned, where blood samples will be taken. The first blood samples will be taken directly before the start of platelet transfusion, the second 1 hour after the end of the platelet transfusion and the third after 24 hours.

Untreated citrate and EDTA blood samples from Visit 1 will be serving as baseline for the coagulation testing. Further citrate blood samples from the first visit will be spiked with different concentrations of fibrinogen in vitro. Untreated citrate and EDTA blood samples will be taken 1 hour and 24 hours after platelet transfusion for comparison. Further citrate blood samples will be spiked with different concentrations of fibrinogen in vitro again 1 hour after platelet transfusion. In addition, randomly chosen samples will be analyzed using confocal microscopy. Routine coagulation analysis include activated partial thromboplastin time (aPTT), prothrombin time(PT), fibrinogen, blood coagulation factor thirteen (FXIII), thromboelastometry (ExTEM & FibTEM) before and after platelet transfusion.

ELIGIBILITY:
Inclusion Criteria:

* patient with the clinical need for platelet transfusion
* age: 18 - 85 years

Exclusion Criteria:

* pregnant or nursing women
* patients who disagree to participate in the study

  * for emergency patients: patients with known refusal of a participation in this clinical trial
* active participation in a clinical trial
* any condition, including the presence of laboratory abnormalities, which would place confound in the ability to interpret data from the study
* any serious medical condition, laboratory abnormalities, or psychiatric illness, that would prevent the subject from signing the informed consent form

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
difference in A30 (ExTEM®) between blood samples after in vitro spiking and compared to those blood samples obtained from the same patients after platelet transfusion | 1 hour after platelet transfusion

SECONDARY OUTCOMES:
Assessment of the difference in the response profile of Blood cell count (EDTA blood sample) | before and 1 hour after platelet transfusion
Standard coagulation tests as aPTT, PT, fibrinogen and FXIII | before and 1 hour after platelet transfusion
Further bleeding management system(ROTEM®)parameters | before and one hour after platelet transfusion
  maximum clot firmness(MCF) clotting time(CT) clot formation time (CFT) lysis index 30 minutes after CT (L30)

CONTACTS AND LOCATIONS:
Overall Officials: Dietmar Fries, Univ-Prof.Dr, Principal Investigator — General and Surgical Intensive Care Medicine, Medical University Innsbruck
Locations (5):
- Austria (3):
  - Central Institution for Blood Transfution and Immunology, Innsbruck, Tyrol
  - Department for Anesthesia and Intensive Care Medicine, Innsbruck, Tyrol
  - General and Surgical Intensive Care Medicine, Innsbruck, Tyrol
- Denmark (2):
  - Faculty of Health Sciences, Centre for Haemophilia and Thrombosis, Aarhus University Hospital, Aarhus, Skejby
  - Faculty of Health Sciences, Department for Anaesthesia and Critical Care Medicine, Aarhus, Skejby